CLINICAL TRIAL: NCT03947814
Title: A Phase 1, Open-label, Single-dose, Parallel-group Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of Pimodivir in Adult Subjects
Brief Title: A Study of Orally Administered Pimodivir in Adult Participants With Renal Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study 63623872FLZ1014 was terminated early based on a strategic business decision by Janssen to end the clinical development program of JNJ-63623872.
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108616; 63623872FLZ1014 (Other: Janssen-Cilag International NV); 2018-002818-12 (EudraCT Number)
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Kidney Failure, Chronic
Keywords: Pimodivir,; JNJ-63623872,; Pharmacokinetics,; Renal impairment,; Kidney disease
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency; Kidney Diseases | interventions — pimodivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: Normal renal function (control group) (Experimental): Participants with normal renal function (glomerular filtration rate [GFR] greater than or equal to [>=] 90 milliliters per minute [mL/min]) will receive single oral dose of 600 mg pimodivir as 2*300 mg tablets.
  Interventions: Drug: Pimodivir
- Part A: Severe renal impairment or ESRD (Experimental): Participants with severe renal impairment (GFR >=15 to less than [<]30 mL/min) who are not on dialysis or end stage renal disease (ESRD) (GFR <15 mL/min) not yet on dialysis will receive single oral dose of 600 mg pimodivir as 2*300 mg tablets.
  Interventions: Drug: Pimodivir
- Part B (Optional): Mild renal impairment (Experimental): Participants with mild renal impairment (GFR >=60 mL/min to <90 mL/min) will receive single oral dose of 600 mg pimodivir as 2*300 mg tablets.
  Interventions: Drug: Pimodivir
- Part B (Optional): Moderate renal impairment (Experimental): Participants with moderate renal impairment (GFR >=30 to <60 mL/min) will receive single oral dose of 600 mg pimodivir as 2*300 mg tablets.
  Interventions: Drug: Pimodivir

INTERVENTIONS:
Drug: Pimodivir — Participants will receive single oral dose of 600 mg pimodivir as 2*300 mg tablets.
  Other Names: JNJ-63623872

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of pimodivir after a single oral dose of 600 milligrams (mg) in adult participants with severe renal impairment who are not on dialysis and in adult participants with end-stage renal disease (ESRD) who are not yet on dialysis compared to adult participants with normal renal function (Part A). Optionally, to evaluate the PK in adult participants with mild and/or moderate renal impairment compared to adult participants with normal renal function (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (Body Mass Index [BMI]; body weight (Kilograms per height^2 [kg/m^2]) between 18.0 and 38.0 kg/m^2, inclusive, and body weight not less than 50 kg, inclusive, at screening
* Participants with normal renal function must have normal values for alanine aminotransferase (ALT) and aspartate aminotransferase (AST) (less than or equal to [<=]1.5*upper limit of laboratory normal range [ULN]) at screening and Day -1 and participants with renal impairment and end-stage renal disease (ESRD) must have values for ALT and AST <=3.0*ULN at screening and Day -1
* Participants with normal renal function must have glomerular filtration rate (GFR) greater than or equal to (>=) 90 milliliters per minute (mL/min) and participants with renal impairment (mild, moderate and severe) and ESRD must have >=60 mL/min to <90 mL/min (for Mild renal impairment); >=30 to <60 mL/min (for Moderate renal impairment); >=15 mL/min to <30 mL/min (for Severe renal impairment not on dialysis); and <15 mL/min (for ESRD not on dialysis)
* Participants with normal renal function must have a systolic blood pressure (after the participant is supine for 5 minutes) between 90 millimeters of mercury (mmHg), extremes included, and diastolic blood pressure no higher than 90 mmHg and participants with renal impairment (mild, moderate and severe) and ESRD must have a systolic blood pressure (after the participant is supine for 5 minutes) between 90 and 159 mmHg, extremes included, and diastolic blood pressure no higher than 99 mmHg. If blood pressure is out of range, 1 repeated assessment is permitted after an additional 5 minutes of rest
* A woman, except if postmenopausal, must have a negative highly sensitive serum pregnancy test (beta human chorionic gonadotropin [beta hCG]) at screening and a negative urine pregnancy test on Day -1

Exclusion Criteria:

* Participant has any surgical or medical condition that potentially may alter the absorption, metabolism, or excretion of the study drug (for example [e.g.], Crohn's disease), with the exception of renal impairment
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody or any other clinically active liver disease at screening
* Participant has a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillin, or drug allergy diagnosed in previous studies with experimental drugs
* Participant has known allergies, hypersensitivity, or intolerance to pimodivir or its excipients
* Participant has evidence of an active infection

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Maximum Observed concentration (Cmax) of Pimodivir | Predose (Day 1), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, and 120 hours postdose on Day 6
  Cmax is the maximum observed concentration.
Area Under Curve From Time of Dosing to the Time of the last Measurable Concentration (AUC[0-last]) of Pimodivir | Predose (Day 1), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, and 120 hours postdose on Day 6
  AUC(0-last) is the AUC from time of dosing to the time of the last measurable (non-below quantification limit) concentration, calculated by linear-linear trapezoidal summation.
AUC from time of dosing to infinity (AUC[0-infinity]) of Pimodivir | Predose (Day 1), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, and 120 hours postdose on Day 6
  AUC(0-infinity) is the AUC from time of dosing to infinity, calculated as AUC(0-last) + Clast/ (lambda[z]), where Clast is the last observed measurable concentration and lambda(z) is the apparent terminal elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 42 (+/-) 2 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (2):
- Germany (2):
  - CRS Clinical Research Services Kiel GmbH, Kiel
  - APEX GmbH, München

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency